CLINICAL TRIAL: NCT06920251
Title: Optimal Infection Prophylaxis Strategy for Relapsed/Refractory Multiple Myeloma Patients Undergoing Elranatamab Therapy
Brief Title: Phase II Trials of Letermovir Prophylaxis in Patients With RRMM Undergoing Elranatamab Therapy
Acronym: OPTIMUS-EL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, JaMin Byun, Professor, MD, PhD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-2503-044-1261
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Relapsed Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Multiple Myeloma | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): This is an experimental cohort designed to evaluate the effectiveness of letermovir in reducing CMV infection in patients with relapsed or refractory multiple myeloma (RRMM) undergoing Elranatamab treatment. Letermovir is administered from Cycle 1 Day 15 (Week 3) to Cycle 4 (Week 16), for a total duration of 98 days.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Elranatamab: Participants will receive SC administration of elranatamab QW, Q2W or Q4W. The initial doses of elranatamab will be 12 mg (C1D1) and 32 mg (C1D4) and will serve as the 2 step-up priming regimen.
  Dexamethasone: Dexamethasone is administered at the dose of 20 mg/day on C1D1, C1D4 and C1D8 as a premedication for elranatamab
  Letermovir: Letermovir is administered at the dose of 480mg/day PO from C1D15 (W3) to C4 (W16) (total of 98 days).
  Other Names: Elranatamab

SUMMARY:
This is an open-label, single arm, multicenter study to evaluate the efficacy of letermovir in the prevention of clinically significant CMV infection in adult, CMV-seropositive relapsed/refractory MM patients undergoing BsAbs therapy.

DETAILED DESCRIPTION:
This is an open-label, single arm, multicenter study to evaluate the efficacy of letermovir in the prevention of clinically significant cytomegalovirus (CMV) infection in adult, CMV-seropositive relapsed/refractory multiple myeloma (MM) patients undergoing Elranatamab therapy.

Elranatamab is bispecific antibody (BsAb), and as BsAbs prolong survivals of MM patients, supportive care is becoming increasingly important to ensure good quality of life and sustain treatment response. Infection control constitutes a major pillar of such supportive care. BsAbs are already very expensive, thus dealing with complications secondary to desultory use will ultimately tantamount to significant financial burden in any given healthcare system. Therefore, implementing risk adaptive prophylactic measures and establishing active monitoring know-hows is important.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  * Subject is ≥ 19 years of age at the time of signing the informed consent form (ICF).

    * Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.

      * Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

        ④ Subjects have documented seropositivity for CMV (CMV IgG seropositvity) at any point. CMV IgG status will be re-checked during screening.

        ⑤ Subject has documented diagnosis of MM and measurable disease, defined as any of the following: A. M-protein ≥ 0.5 g/dL by serum protein electrophoresis (sPEP) or B. M-protein ≥ 200 mg/24-hour urine collection by urine protein electrophoresis (uPEP) or C. For subjects without measurable disease in sPEP or uPEP: serum free light chain (sFLC) levels > 100 mg/L (10 mg/dL) involved light chain and an abnormal kappa/lambda FLC ratio.

        *Patients with extramedullary disease (EMD) only will be allowed to participate if there is a measurable extramedullary lesion. These patients require PET-CT follow-up for response evaluation.

        ⑥ Subject has received 3 or more prior lines of antimyeloma therapy. (Note: One line can contain several phases [e.g., induction, (with or without) hematopoietic stem cell transplant, (with or without) consolidation, and/or (with or without) maintenance therapy).

        ⑦ Subject must have received at least one proteasome inhibitor, one immunomodulatory drug, and one anti-CD38 antibody.
        * Subject must have documented disease progression during or after their last antimyeloma regimen.

          * Subject has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.

            * Individual of childbearing potential (IOCBP) must:

A. Have two negative pregnancy tests as verified by the investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.

B. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, 2 forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting study treatment, during the study treatment (including dose interruptions), and for at least 90 days after the last dose of letermovir or 4 months after the last dose of elranatamab, whichever is longer.

⑪ Male subjects must: A. Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant individual or an individual of childbearing potential while participating in the study, during dose interruptions and for at least 90 days after the last dose of letermovir, even if he has undergone a successful vasectomy.

* True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

  * Male subjects must agree to refrain from donating sperm while on study treatment, during dose interruptions and for at least 90 days following last dose of letermovir.

    * Females must agree to refrain from donating eggs while on study treatment and for at least 90 days after last dose of letermovir.

      * Subjects must agree to refrain from receiving live vaccines while on study treatment, during dose interruptions and for at least 90 days following the last dose of elranatamab.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Subject who has a history of CMV end-oragn disease within 6 months prior to enrollment.
  2. Subject who has evidence of CMV viremia at screening (D-7 CMV DNA results required - for specifics refer to section 5.3 and schedule of activities; SoA).
  3. Subject who has received within 7 days prior to screening or plans to receive during the study ant of the following:

     A. Ganciclovir B. Valganciclovir C. Foscarnet D. Acyclovir, at doses > 3200mg PO per day or > 25mg/kg IV per day E. Valacyclovir, at doses > 3000mg PO per day F. Famciclovir, at doses > 1500mg PO per day
  4. Subject who has suspected or known hypersensitivity to active or inactive ingredients of letermovir formulations.
  5. Subject has received any of the following. A. Plasmapheresis within the last 28 days of initiating study treatment B. Major surgery (as defined by the investigator) within 28 days of initiating study treatment.
  6. Subject has previously received allogeneic stem cell transplantation within a year during prior therapy or received autologous stem cell transplantation within 12 weeks of initiating study treatment. Patients who received allogeneic stem cell transplantation should not have evidence of active graft-versus-host disease (GVHD) and off any immunosuppressants.
  7. Subject has plasma cell leukemia defined by IMWG definition for primary plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or clinically significant light-chain amyloidosis.
  8. Subject with known central nervous system (CNS) involvement with myeloma.
  9. Subject has any significant medical condition, including active or uncontrolled infection, presence of laboratory abnormality, or psychiatric illness that places the subject at an unacceptable risk for treatment-related complications, if he/she were to participate in the study.
  10. Coronavirus disease 2019 (COVID-19) within 7 days for mild or asymptomatic infections or 14 days for moderate/severe infections prior to initiating study intervention. A longer duration may be needed based on the investigator's clinical judgment.

      A. Acute symptoms must have resolved and there are no sequelae that would place the participant at a higher risk of receiving study intervention, based on investigator assessment. No repeat/follow-up COVID-19 testing is required.
  11. Subject has any condition that confounds the ability to interpret data from the study.
  12. Subject has any of the following laboratory abnormalities:

      A. Absolute neutrophil count (ANC) < 1,000/µL. B. Platelet count < 25,000/µL. C. Estimated glomerular filtration rate (eGFR) < 30 mL/min or requiring dialysis. eGFR will be calculated using the Modification of Diet in Renal Disease (MDRD) formula.

      D. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN) E. Serum total bilirubin > 1.5 × ULN, or for participants with documented Gilbert's syndrome > 3.0 mg/dL
  13. Subject with gastrointestinal disease or surgery (e.g., gastric bypass surgery) that may significantly alter the absorption of letermovir and/or other oral study treatment.
  14. Subject has a prior history of malignancies other than MM, except if the participant has been free of the disease for ≥ 3 years. Patients with CIS treated with curative intent are not excluded if less than 3 years. Exceptions would include basal cell and squamous cell cancer of the skin treated with curative intent.
  15. Subject has received immunosuppressive medication within the last 14 days of initiating study treatment. The following are exceptions to this criterion: a. Intranasal, inhaled, topical or local corticosteroid injections (e.g., intra-articular injection). b. Systemic corticosteroids at doses that do not exceed 10 mg/day of prednisone or the equivalent. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
  16. Impaired cardiovascular function or clinically significant cardiovascular diseases, defined as any of the following within 6 months prior to enrollment:

      A. Acute myocardial infarction or acute coronary syndromes (eg, unstable angina, coronary artery bypass graft, coronary angioplasty or stenting, symptomatic pericardial effusion); B. Clinically significant cardiac arrhythmias (eg, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia); C. Thromboembolic or cerebrovascular events (eg, transient ischemic attack, cerebrovascular accident, deep vein thrombosis [unless associated with a central venous access complication] or pulmonary embolism); D. Prolonged QT syndrome (or QTcF >470 msec at screening); E. LVEF < 40% as determined by a MUGA scan or echocardiography.
  17. Subject has uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.
  18. Subject who has had a live vaccine within 3 months of start of study therapy.
  19. Subject is positive for human immunodeficiency virus (HIV), chronic or active hepatitis B, active hepatitis A, or active hepatitis C:

      A. Known positive HIV status. B. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] either acute or chronic hepatitis). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBcAb] and/or antibodies to hepatitis B surface antigen [anti-HBsAb]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded.

      EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.

      EXCEPTION: Subjects with positive anti-HBcAb but negative HBsAg and negative anti-HBsAb profiles are eligible if HBV DNA PCR is negative.

      C. Known to be seropositive for hepatitis C virus (HCV); anti-HCV antibody positive and HCV- ribonucleic acid (RNA) quantitation positive.
  20. Ongoing Grade 3 or higher peripheral sensory or motor neuropathy, history of Guillan-Barre syndrome (GBS) or GBS variants, or history of any Grade >3 peripheral motor polyneuropathy.
  21. Subject is an individual who is pregnant, nursing or breastfeeding, or who intends to become pregnant during participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with clinically significant CMV infection during 6 cycles of elranatamab treatment | From Cycle 1 Day 1 to completion of Cycle 6 (Week 24; each cycle is 28 days)
  Clinically significant CMV infection is defined as the occurrence of either one of the following outcomes:
  1. onset of CMV end-organ disease or
  2. initiation of anti-CMV pre-emptive therapy based on documented CMV viremia* and the clinical condition of the subject. Initiation of pre-emptive therapy refers to the practice of initiating therapy with the following approved anti-CMV agents when active CMV viral replication is documented: ganciclovir, valganciclovir, foscarnet, and/or cidofovir.
     * Viral load threshold for initiating pre-emptive therapy is viral DNA ≥ 500 IU/mL in 2 consecutive assessments separated by at least 1 day, or, single viral DNA ≥ 1,000 IU/mL

SECONDARY OUTCOMES:
Proportion of subjects with clinically significant CMV infection during 12 cycles of elranatamab treatment | From Cycle 1 Day 1 to completion of Cycle 12 (each cycle is 28 days)
  Clinically significant CMV infection is defined as the occurrence of either one of the following outcomes:
  1. onset of CMV end-organ disease or
  2. initiation of anti-CMV pre-emptive therapy based on documented CMV viremia* and the clinical condition of the subject. Initiation of pre-emptive therapy refers to the practice of initiating therapy with the following approved anti-CMV agents when active CMV viral replication is documented: ganciclovir, valganciclovir, foscarnet, and/or cidofovir.
     * Viral load threshold for initiating pre-emptive therapy is viral DNA ≥ 500 IU/mL in 2 consecutive assessments separated by at least 1 day, or, single viral DNA ≥ 1,000 IU/mL
Incidence of CMV disease during the first 6 and 12 cycles of elranatamab | From Cycle 1 Day 1 to completion of Cycle 6 and Cycle 12, respectively (each cycle is 28 days)..
Incidence of CMV viremia during the first 6 and 12 cycles of elranatamab | From Cycle 1 Day 1 to completion of Cycle 6 and Cycle 12, respectively (each cycle is 28 days).
  Virus detection of any titer. CMV viremia refers to CMV DNA levels in the plasma (=CMV DNAemia).
Toxicity | From Cycle 1 Day 1 to study completion, an average of 1 year.
  Type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs to study treatment.
Tolerability | From Cycle 1 Day 1 to study completion, an average of 1 year.
  Study treatment adherence rate, including elranatamab dose and schedule modifications

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided